CLINICAL TRIAL: NCT04682548
Title: Estimating Prevalence of COVID-19 Infection and SARS-CoV-2 Antibodies in MS Patients With and Without Ocrelizumab Treatment, and Comparing Immune Responses to COVID-19 in MS Patients on Ocrelizumab and Healthy Controls
Brief Title: Estimating Prevalence of COVID-19 Infection and SARS-CoV-2 Antibodies in MS Patients
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 20-01799
Record Dates: First submitted 2020-12-22; First posted 2020-12-23 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Multiple Sclerosis; Covid19
Keywords: Disease-Modifying Therapy
MeSH Terms: conditions — Multiple Sclerosis; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be obtained from participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This non-interventional, biospecimen collection study is designed to help us better understand whether MS patients have impaired immune defenses to COVID-19 infection. The potential influence of immune modulating medications for MS will be considered through these exploratory studies. This study is also designed to provide context for interpretation of anti-SARS CoV2 serologies in MS patients during convalescence from COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria (Part A and B):

● Patient is outside of infectious period of COVID-19 defined as follows:

* Patient with mild to moderate illness who are not severely immunocompromised:

  * At least 10 days have passed since symptoms first appeared and
  * At least 24 hours have passed since last fever without the use of fever-reducing medications and
  * Symptoms (e.g. cough, shortness of breath) have improved
* Patient with severe to critical illness or who are severely immunocompromised:

  * At least 10 days and up to 20 days have passed since symptoms first appeared
  * At least 24 hours have passed since last fever without the use of fever-reducing medications and
  * Symptoms (e.g. cough, shortness of breath) have improved

    * Clinician-diagnosed MS treated or untreated with an approved DMT,
    * Ages 18 to 60,
    * EDSS 0 - 7,
    * Able to give informed consent,
    * Able to complete, or have someone help complete the patient questionnaire,
    * No high dose steroids, or IVIG, or PLEX use within 3 months of blood sample,
    * No convalescent plasma and/or polyclonal antibody treatments for COVID-19 within 3 months of blood sample collection.

Inclusion Criteria (Part B only)

* COVID-19 positive patients, who received OCR within 6 months of COVID 19 infection,
* EDSS 0 - 6.

Inclusion Critera (Redraws Only)

* Completed standard of care COVID-19 vaccination series
* On Ocrevus, glatiramer, interferon b, or not on any treatment disease-modifying treatment at the time of vaccination.

Exclusion Criteria (Part A and B):

* Concurrent immunosuppressive therapy, active systemic cancer, primary or acquired immunodeficiency (i.e., CVID, HIV infection),
* Active drug or alcohol abuse,
* Other anti-CD20 therapy apart from OCR,
* Uncontrolled diabetes mellitus,
* End-organ failure (cardiac, pulmonary, renal, hepatic),
* Systemic lupus erythematosus (SLE).

Exclusion Criteria (Part B only):

* EDSS >6,
* Active infection (e.g., hepatitis).

Exclusion Criteria (Healthy Controls Sample)

* Concurrent immunosuppressive therapy, active systemic cancer, primary or acquired immunodeficiency (e.g. CVID, HIV infection),
* Active ongoing drug or alcohol abuse,
* Age >60 or <18,
* Uncontrolled diabetes mellitus,
* End-organ failure (cardiac, pulmonary, renal, hepatic),
* SLE
* No high dose steroids, or intravenous immunoglobulin (IVIG) or plasma exchange (PLEX) use within 3 months of blood sample collection,
* No convalescent plasma and/or polyclonal antibody treatments for COVID-19 within 3 months of blood sample collection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Projected study size is 1000 MS patients for primary objective and additional 40 non-autoimmune COVID-19 convalescent control and 20 COVID-19 negative healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 920 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Seropositivie Rate Against SARS-CoV-2 | Baseline, Day 0
  Seropositivity rate against SARS-CoV-2 (nucleocapsid and/or spike proteins, as available) as measured by the Roche DIA antibody assay in MS patients.

SECONDARY OUTCOMES:
T Cell Response | Baseline, Day 0
  SARS-CoV-2 specific T cells will be measured using a well-validated assay such as ELISpot (enzyme-linked immune absorbent spot) to measure T cell responses to stimulation.

OTHER OUTCOMES:
T Cell response | Baseline, Day 0
  SARS-CoV-2 specific T cells will be measured using a well-validated assay such as ELISpot (enzyme-linked immune absorbent spot) to measure T cell responses to stimulation.
T Cell response | up to week 48 Post-Vaccination
  SARS-CoV-2 specific T cells will be measured using a well-validated assay such as ELISpot (enzyme-linked immune absorbent spot) to measure T cell responses to stimulation.
SARS-CoV-2 Antibodies Level | Baseline, Day 0
  SARS-CoV-2 antibodies will be measured and assessed with Roche DIA Assay
SARS-CoV-2 Antibodies Level | up to week 48 Post-Vaccination
  SARS-CoV-2 antibodies will be measured and assessed with Roche DIA Assay

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Kister, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Curtin R, Velmurugu Y, Dibba F, Hao Y, Sreenivasaiah C, Khodadadi-Jamayran A, Nyovanie S, Kim A, Samanovic ML, Mulligan M, Priest J, Cabatingan M, Winger RC, Patskovsky Y, Kister I, Silverman GJ, Krogsgaard M. Persistent Classical and Atypical Memory B Cells Underlie Heterogeneous Vaccine Responses in Ocrelizumab-Treated Multiple Sclerosis. bioRxiv [Preprint]. 2025 Nov 4:2025.11.03.686372. doi: 10.1101/2025.11.03.686372. PMID 41279857